CLINICAL TRIAL: NCT04513418
Title: Effects of Preoperative Enteral Immunonutrition for Esophageal Cancer Patients Given Neoadjuvant Chemoradiotherapy
Acronym: POINT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hecheng Li M.D., Ph.D (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Zhongshan Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Hecheng Li M.D., Ph.D, Director, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RTS-011
Record Dates: First submitted 2020-08-07; First posted 2020-08-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Neoplasms; Neoadjuvant Therapy; Enteral Nutrition; Nutrition Therapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): Patients receive omega-3 fatty-acid enriched enteral nutritional emulsion during the neoadjuvant chemoradiotherapy. Patients are meanwhile encouraged to intake 25-30kcal/kg through regular food.
  Interventions: Dietary Supplement: Preoperative immunonutrition
- Control group (No Intervention): Patients are encouraged to intake 25-30kcal/kg through regular food without supplemental nutritional support before esophagectomy.

INTERVENTIONS:
Dietary Supplement: Preoperative immunonutrition — Preoperative immunonutrition includes an omega-3 fatty-acid enriched enteral nutritional emulsion given by oral intake, nasogastric feeding tube or jejunostomy 600ml per day, lasting for the whole period of neoadjuvant chemoradiation. Meanwhile, oral intake is encouraged to reach 25-30kcal/kg through regular food.
  Arms: Interventional group

SUMMARY:
This randomized controlled trial will evaluate the effects of preoperative enteral immunonutrition in esophageal cancer patients undergoing neoadjuvant therapy. The purpose of this study is to determine whether preoperative immune-modulating diet before surgery can improve the rate of complications and other perioperative outcomes.

DETAILED DESCRIPTION:
Esophageal cancer ranks the fourth in mortality and the sixth in incidence among cancers in China according to the latest report of cancer epidemiology. Although the development of neoadjuvant therapy and radical esophagectomy have improved the prognosis of esophageal cancer patients, dysphagia and digestive tract reconstruction can cause malnutrition and infection-related complications. Postoperative enteral and parenteral nutrition have proved to be effective in improving outcomes after esophagectomy. However, whether to provide a preoperative nutritional support for patients with resectable esophageal cancer remains controversial.

This prospective randomized controlled trial will evaluate the effects of preoperative enteral immunonutrition in esophageal cancer patients undergoing neoadjuvant therapy. The purpose of this study is to determine whether preoperative immune-modulating diet before surgery can improve the rate of complications and other perioperative outcomes.

The sample size is estimated with the hypothesis that preoperative immunonutrition during the neoadjuvant therapy can reduce postoperative nutrition and immune-related complications after esophagectomy. According to the previously published articles, the required sample size of interventional and control arm (ratio=2:1) was calculated as 137 cases and 69 cases to detect the reduction in related complications from 50% to 30% based on a bilateral significance level (α) of 0.05 and a power of test (1-β) of 0.80. Considering an estimated drop rate of 15%, the minimum sample size of this study is 244 patients, 162 cases in the interventional group and 82 in the control group. After signing the informed consent, every eligible participant will be randomized into either group based on a computer-generated random number. Blinding will not be applied to patients and surgeons due to the difficulty in clinical practice but outcomes assessor will be masked.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal cancer
* Staging as cT2N0M0 with high-risk lesions (lymphovascular invasion, ≥3cm, poorly differentiated) / cT1b-2N+M0 / cT3-4aN0-3M0 with the need of neoadjuvant therapy before radical esophagectomy
* Tolerance with oral intake (at least fluid diet)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Body Mass Index (BMI) ≥ 18.5 kg/m2 before recruitment
* Patient's approval and written informed consent

Exclusion Criteria:

* Expected survival time less than 6 months
* Complete dysphagia
* Pregnant or breast-feeding women
* Unable to obey the interventions because of any reasons
* Serious co-morbidities (cardiac, pulmonary, liver, kidney, brain, hematologic, endocrine and other diseases) in patients who cannot tolerate neoadjuvant therapy and/or surgery
* History of previous thoracic or abdominal surgery
* History of other malignant tumor (previous or current)
* Patients with primary small cell carcinoma of the esophagus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative nutrition and immune-related complications | Up to 30 days after surgery
  Rate of gastrointestinal complications (anastomotic leakage, gastrointestinal dysfunction), metabolic complications (electrolyte disturbances, liver or renal dysfunction) and infectious complications(wound infection, catheter-related infection, pneumonia, sepsis, or other infections requiring antibiotics).

SECONDARY OUTCOMES:
Completion rate of neoadjuvant therapy and esophagectomy | 2-3 months before surgery
Adverse events during neoadjuvant chemoradiotherapy | 2-3 months before surgery
Pathological complete response rate (pCR) | 2-3 months before surgery
Blood loss | At operation day
Duration of surgery | At operation day
Rate of surgery-related complications | At operation day
  Conversion to open surgery, recurrent nerve injury, cardiac and cerebrovascular accident
Length of hospital stay | Postoperative in-hospital stay
Hospitalization costs | Postoperative in-hospital stay
30-day and 90-day mortality | Up to 90 days after surgery
Weight loss | From neoadjuvant chemoradiotherapy to 6 months after surgery
Change in PG-SGA score after surgery | From neoadjuvant chemoradiotherapy to 6 months after surgery
Change in biochemical indicators after surgery | From neoadjuvant chemoradiotherapy to 6 months after surgery
  WBC, hemoglobin, albumin, CRP, TNF-α, interleukins, IgA, IgG, IgM, fasting blood-glucose
Score of EORTC QLQ-C30 and OES-18 scale | 1-year, 3-year, and 5-year after surgery
  Quality of life
Long-term survival | 1-year, 3-year, and 5-year after surgery
  Overall survival (OS) and progression-free survival (PFS)

OTHER OUTCOMES:
Minimal residual disease (MRD) | Before and after neoadjuvant chemoradiotherapy, 7-14 days after surgery
  Studies suggest that MRD monitoring through circulating tumor DNA (ctDNA) can predict whether a patient has achieved pCR after neoadjuvant chemoradiotherapy, thereby evaluating the efficacy of the treatment. Therefore, in order to explore whether enteral immunonutrition influences the efficacy of neoadjuvant chemoradiotherapy, we added the exploratory endpoint of MRD detection.
Microbiomics analysis | 1 week before neoadjuvant chemoradiotherapy, 2-3 days before surgery
  By collecting fecal samples before and after neoadjuvant chemoradiotherapy and utilizing metagenomic sequencing, we aim to investigate the impact of enteral immunonutrition on the gut microbiome distribution in patients with esophageal cancer.
Metabolomic analysis | 1 week before neoadjuvant chemoradiotherapy, 2-3 days before surgery
  By collecting peripheral blood samples before and after neoadjuvant chemoradiotherapy and utilizing mass spectrometry, we aim to investigate the impact of enteral immunonutrition on the metabolomic distribution in patients with esophageal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, PhD, MD, Principal Investigator — Ruijin Hospital
Locations (6):
- China (6):
  - Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Cancer Hospital of University of Chinese Academy of Sciences, Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao Y, Han D, Yang S, Shi Y, Zhao S, Jin Q, Li J, Li C, Zhang Y, Shen W, He J, Wang M, Ji G, Li Z, He Y, Chen Q, Wei W, Chen C, Gong X, Wang J, Tan L, Wang H, Li H. Effects of pre-operative enteral immunonutrition for esophageal cancer patients treated with neoadjuvant chemoradiotherapy: protocol for a multicenter randomized controlled trial (point trial, pre-operative immunonutrition therapy). BMC Cancer. 2022 Jun 13;22(1):650. doi: 10.1186/s12885-022-09721-y. PMID 35698100